CLINICAL TRIAL: NCT05776251
Title: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) for Persistent Symptoms From Lyme Disease: a Feasibility, Tolerability, and Safety Study
Brief Title: taVNS for Persistent Symptoms From Lyme Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Brian A Fallon, Professor of Clinical Psychiatry, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV3947
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Post-Treatment Lyme Disease
Keywords: Lyme Disease; Vagus Nerve Stimulation; taVNS; Fatigue
MeSH Terms: conditions — Post-Lyme Disease Syndrome; Lyme Disease; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PTLD - active taVNS (Experimental): Participants with Post-treatment Lyme Disease (PTLD) will start with 40 sessions (i.e., 4 weeks of Monday to Friday, twice daily treatments that last 1 hour each session) to receive transcutaneous auricular Vagus Nerve Stimulation (taVNS). If compliance is less than 70% in at least 3 of the first 4 open label treated participants, then the investigators will modify the treatment design accordingly.
  Interventions: Device: taVNS

INTERVENTIONS:
Device: taVNS — Includes the use of Soterix Medical Device, which consists of a handheld "smart-phone" size device. There are two electrodes (designed for studies in infants) with small patches that the participant places on the external ear (the cymbals conchae and the tragus). The stimulation intensity is personalized for each participant based on perceptual threshold.

SUMMARY:
This study is one of the first studies to investigate a non-antibiotic approach to the treatment of symptoms that persist after antibiotic treatment for Lyme disease (PTLS). Transcutaneous auricular vagus nerve stimulation (taVNS) offers the potential of being an effective and non-toxic approach to reduce the burden of multisystem symptoms in patients with PTLS. This study seeks to address an important goal: to assess the safety, feasibility, and tolerability of a new non-invasive, non-pharmacologic treatment for patients with symptoms that persist despite prior antibiotic treatment for Lyme disease.

DETAILED DESCRIPTION:
Musculoskeletal pain, fatigue, and cognitive and mood problems are common persistent disabling symptoms among individuals with post-treatment Lyme Disease. Each year in the United States, approximately 476,000 individuals are newly diagnosed with Lyme disease and 10-20% of these go on to have persistent or relapsing symptoms that are not responding to the current best antibiotic therapies.

Individuals with persistent infection are likely to respond best to additional antibiotic therapy. Individuals with post- infectious causes require other approaches - such as ones that impact ongoing inflammation or altered neural circuits and metabolism. Safe and effective treatment for these individuals with persistent symptoms represents a prominent unmet need.

Vagus nerve stimulation (VNS) may be a treatment with considerable impact for patients with post-treatment Lyme disease. The vagus nerve (the 10th and longest cranial nerve) impacts the central nervous system, the autonomic nervous system (e.g, heart, lungs, digestive tract), and the systemic inflammatory response. It has also been shown to play a role in cognition, pain, mood disorders, inflammation, and immune function. Research over the last 2 decades has demonstrated that electrical stimulation of the vagus nerve can have multiple salutary effects in both animal models of disease and human illness. Until very recently, VNS has been considered an invasive intervention, reserved for patients with refractory disease, as it requires surgery to implant the device; this approach is costly and puts patients at risk of infection and other complications. These factors have limited the accessibility and broad application of VNS. A non-invasive approach to VNS would increase affordability, accessibility, and decrease risk. This is now possible. The first non-invasive external VNS device was cleared by the FDA for the treatment of cluster headaches and migraines in 2017.

ELIGIBILITY:
Inclusion Criteria:

* History of either Definite or Highly Probable Past Lyme disease diagnosed and treated by a health care provider more than 6 months previously.
* Have one or more current symptoms attributed to Lyme disease that were also present during the initial 6-month period after diagnosis and antibiotic treatment of Lyme disease.
* Individuals reporting that current symptoms cause clinically significant distress or impairment in functioning.
* Previously treated for Lyme disease with at least two courses of antibiotics considered appropriate for Lyme disease.
* Individuals who agree to not start a new medical or psychiatric treatment (that might impact study outcomes) for their chronic symptoms during the course of this study (unless deemed necessary by their primary care physician (PCP)).
* Individuals whose current treatment (that might impact study outcomes) has been stable for at least 6 weeks prior to baseline visit.
* Lives in the U.S. and owns a smartphone, tablet or computer with Internet access.
* Able to read and understand English to be able to provide informed consent.
* Able and willing to come to Columbia University Irving Medical Center in NYC for 3-5 study visits.
* Willingness to have a 12-lead electrocardiogram (EKG) when evaluated on site and, if an EKG was conducted in the past year, willingness to try to obtain that EKG for us to review.
* Current moderate to severe fatigue. At least moderate intensity at study screening (a score of 4 or more on the Fatigue Severity Scale (FSS)).
* Ability to allocate sufficient time for the treatment sessions, including 6 sessions that will be monitored during work hours (8 am to 6 pm).

Exclusion Criteria:

* Current or past history of cardiovascular disorder(s) (coronary artery disease, peripheral artery disease, stroke, aortic disease, or other major cardiac condition). A history within the last year of unexplained fainting spells or of vasovagal syncope or feeling faint in response to medical settings or pain. Symptomatic bradycardia, orthostatic (postural) hypotension not correctable by fluid intake (i.e., a drop of >20 mm Hg systolic, 10 mm Hg diastolic or both), or persistent hypotension (BP below 90 mmHg systolic).
* Abnormal EKG findings (e.g., significant bradycardia) considered significant by a cardiologist.
* A diagnosed current major central nervous system disease (e.g., multiple sclerosis (MS), epilepsy, neurodegenerative diseases, ischemic stroke, Parkinson's, traumatic brain injury with cognitive impairment, etc.) or a history of brain surgery or brain tumors.
* A current psychiatric disorder that might impact treatment compliance (e.g., bipolar disorder, psychosis, substance abuse).
* Suicidal ideation with method, plan or intent in the last 6 months or a lifetime history of suicidal behavior.
* Current moderate-severe or severe depression (T-score of 65 or higher on the PROMIS-Emotional Distress-Depression SF) at screening.
* Current serious unstable medical illness.
* Currently taking opiate-based medication or have taken antibiotics in the last 6 weeks for tick-borne illness.
* Ear-related: a) facial or ear pain; b) recent ear trauma; c) damage to left or right ear or anatomy that does not allow taVNS; d) ear infection (otitis media or externa); e) scar or inflammation on ear; f) Cochlear implants.
* Currently or recently (within 6 months) in a clinical trial of an investigational medicinal product or another medical device.
* Females who are pregnant or planning to become pregnant during the course of this study.
* Unable to connect to the Internet during treatment phase.
* Individuals with an active external or implanted electrical medical device (e.g., cardiac pacemaker, hearing aid implant) or any metal implant above the level of the neck.
* Individuals who have had surgery to cut the vagus nerve in the neck (cervical vagotomy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Up to 4 weeks
  To assess feasibility of conducting a study of taVNS for patients with persistent symptoms after Lyme disease, recruitment will be calculated from the number of participants in the study.
Compliance Rate | Up to 4 weeks
  To assess feasibility of taVNS for patients with persistent symptoms after Lyme disease, compliance will be measured as the number of completed sessions per participant.
Drop-out Rate | Up to 4 weeks
  To assess tolerance to taVNS, the drop-out rate will be calculated from the number of participants who discontinue from the study.
Ratings of Treatment Satisfaction (Likert Scale) | Up to 4 weeks
  To assess tolerance to taVNS, participants will be asked to rate their satisfaction with the treatment experience on a Likert Scale, with 1 (min) indicating "very dissatisfied" to 5 (max), indicating "very satisfied". A higher score indicates a better outcome.
Total Number of Treatment Emergent Adverse Events | Up to 4 weeks
  To assess safety of taVNS, the total number of treatment emergent adverse events will be assessed using the Systematic Assessment for Treatment Emergent Effects (SAFTEE) tool.

CONTACTS AND LOCATIONS:
Overall Officials: Brian A. Fallon, MD, Principal Investigator — Columbia University
Locations (1):
- Lyme and Tick-Borne Diseases Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Homepage for Columbia University's Lyme and Tick-Borne Diseases Research Center — http://columbia-lyme.org